CLINICAL TRIAL: NCT07360665
Title: PEP - Physical Exercise for Psychosis: A Study Protocol
Brief Title: Multimodal Physical Exercise Program (Physical Exercise for Psychosis) for People With Psychosis Treated With Long-Acting Injectable Antipsychotics
Acronym: PEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trás-os-Montes and Alto Douro (Other)
Collaborators: Centro Hospitalar De Trás-Os-Montes E Alto Douro, E.P.E. (Unknown)
Responsible Party: Principal Investigator, Sofia Silva, Principal Investigator, University of Trás-os-Montes and Alto Douro
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024.04489.BDANA; CES REG. 1612 (Other: Ethics Committee, Local Health Unit of Trás-os-Montes and Alto Douro, Vila Real, Portugal)
Record Dates: First submitted 2025-12-17; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Psychotic Disorders; Schizophrenia Spectrum Disorders (SSD); Severe Mental Illness
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients diagnosed with psychosis who are receiving farmacological treatment and exercise program. (Experimental): Patients aged 18 years or older, diagnosed with psychosis, undergoing treatment with LAIs, and holding a certificate of autonomy issued by their psychiatrist, with the additional requirement for the experimental group to reside near the location of the physical exercise sessions.
  Interventions: Other: Physical Exercise
- Patients diagnosed with psychosis who are receiving farmacological treatment. (No Intervention): Patients aged 18 years or older, diagnosed with psychosis, undergoing treatment with LAIs, and holding a certificate of autonomy issued by their psychiatrist.

INTERVENTIONS:
Other: Physical Exercise — The program will be multimodal, integrating various exercise components. The aerobic component will consist of activities like walking, cycling, and circuit training. The functional strength component will include 2 to 3 exercises for the lower limbs, 2 to 3 exercises for the upper limbs, 1 to 2 exercises for the trunk and abdominal muscles, as well as 1 to 2 multi-joint exercises like burpees, swing kettlebell, among others. Lastly, the program will also incorporate mobility, balance, and flexibility exercises, such as stretching, postures, and joint mobilization.
  Other Names: Multimodal Physical Exercise
  Arms: Patients diagnosed with psychosis who are receiving farmacological treatment and exercise program.

SUMMARY:
People with psychotic disorders, such as schizophrenia, often experience significant difficulties in daily functioning, physical health, and quality of life. Long-acting injectable antipsychotics are an important part of treatment, but they can be associated with metabolic side effects and reduced physical fitness. Physical exercise has shown potential benefits for mental and physical health in this population; however, structured exercise programs implemented in real-world psychiatric services are still limited.

The purpose of this study is to evaluate the feasibility and clinical impact of a structured, multimodal physical exercise program for adults with psychosis who are receiving long-acting injectable antipsychotic treatment. The study aims to determine whether participation in a supervised exercise program can improve physical functioning, psychological well-being, and selected biological markers related to brain health and metabolism.

This study will be conducted in an outpatient psychiatric setting in Portugal and will include adults diagnosed with psychosis who are currently treated with long-acting injectable antipsychotics. Participants will be allocated to either an exercise group or a control group receiving usual care. The exercise program will last 24 weeks and will include aerobic, strength, mobility, and flexibility exercises, with supervised sessions conducted by qualified professionals.

Participants will be assessed at baseline, during the intervention, after completion of the program, and at follow-up. Assessments will include measures of physical function, body composition, psychological well-being, quality of life, and blood-based biomarkers such as brain-derived neurotrophic factor, dopamine, serotonin, and metabolic indicators.

The main hypothesis of this study is that individuals who participate in the physical exercise program will show improvements in physical function, mood, and overall well-being compared with those receiving usual care alone. The results of this study are expected to provide practical evidence to support the integration of structured physical exercise as an adjunct to routine psychiatric care for people with psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Clinical diagnosis of psychosis;
* Currently undergoing treatment with long-acting injectable antipsychotics (LAIs);
* Follow-up at the Antipsychotic Clinic of ULSTMAD;
* Certificate of autonomy issued by the treating psychiatrist, confirming the participant's capacity to engage in the study procedures;
* Ability to provide written informed consent, either personally or through a legal representative;
* (Experimental group only) Residence within a reasonable distance from the physical exercise intervention site to allow attendance at supervised sessions.

Exclusion Criteria:

* Attendance below 85% of the supervised exercise sessions (experimental group);
* Failure to complete the four main assessment time points;
* Withdrawal or lack of informed consent at any stage of the study;
* Not prescribed long-acting injectable antipsychotics (LAIs);
* Not affiliated with or followed at the Antipsychotic Clinic of ULSTMAD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Body mass/weight | Baseline, 12 weeks, 24 weeks, 8-week post-intervention follow-up
  Body mass/weight measured in kilograms using a calibrated scale.
Body mass index (BMI) | Baseline, 12 weeks, 24 weeks, 8-week post-intervention follow-up
  BMI calculated as weight (kg) / height (m²)
Body fat percentage | Baseline, 12 weeks, 24 weeks, 8-week post-intervention follow-up
  Body fat percentage assessed by electrical bioimpedance analysis
Lean body mass | Baseline, 12 weeks, 24 weeks, 8-week post-intervention follow-up
  Lean body mass (kg) assessed by electrical bioimpedance analysis
Sit-to-Stand Test _ 30s | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  Used to measure lower limb strength and endurance through the number of repetitions performed in a specific period.
Handgrip Test | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  Used to assess upper limb muscle strength
European Health Interview Survey - Quality of Life 8-item Index (EUROHIS-QOL-8) | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  The European Health Interview Survey - Quality of Life 8-item Index (EUROHIS-QOL-8) is an 8-item self-report questionnaire assessing overall quality of life across physical, psychological, social, and environmental domains. Each item is rated on a 5-point Likert scale, resulting in a total score ranging from 8 to 40. Higher total scores indicate better perceived quality of life. The scale demonstrates good psychometric properties and is suitable for use in clinical and research settings.
Patient Health Questionnaire-9 - PHQ-9 | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-administered questionnaire designed to assess the severity of depressive symptoms based on the diagnostic criteria for major depressive episodes. Each item is scored on a 4-point Likert scale (0-3), yielding a total score ranging from 0 to 27. Higher total scores indicate greater severity of depressive symptoms. The PHQ-9 is widely used in clinical and research settings and demonstrates good psychometric properties.
Positive and Negative Affect Scale (PANAS) | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  The Positive and Negative Affect Schedule (PANAS) is a 20-item self-report questionnaire designed to assess affective states, comprising two independent 10-item subscales: Positive Affect (PANAS-PA) and Negative Affect (PANAS-NA). Each item is rated on a 5-point Likert scale (1-5), yielding subscale scores ranging from 10 to 50. Higher scores on the Positive Affect subscale indicate higher levels of positive affect, whereas higher scores on the Negative Affect subscale indicate higher levels of negative affect. The PANAS is widely used in clinical and research settings and demonstrates good psychometric properties.
Serum Brain-Derived Neurotrophic Factor (BDNF) levels | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  Serum BDNF concentration quantified using standardized Human BDNF ELISA Kit (Abcam). BDNF is a key neurotrophic marker associated with neuroplasticity and treatment-related neurobiological adaptations. Units: ng/mL.
Serum lipid profile | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  Assessment of serum lipid parameters including total cholesterol, HDL cholesterol, LDL cholesterol (direct or calculated), and triglycerides, according to hospital laboratory reference standards. Units: mg/dL.
  Hospital laboratory references:
  * Total cholesterol: < 200 mg/dL
  * LDL cholesterol: < 130 mg/dL
  * HDL cholesterol: > 60 mg/dL
  * Triglycerides: < 150 mg/dL
Glycemic and metabolic markers | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  Evaluation of fasting blood glucose and glycated hemoglobin (HbA1c) as indicators of glycemic control and metabolic health.
  Units:
  * Glucose: mg/dL
  * HbA1c: %
  Hospital reference values:
  * Glucose: 74-106 mg/dL
  * HbA1c: 4.0-6.0 %
Serum Serotonin levels | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  Quantification of serotonin concentration in serum using standardized laboratory procedures. Higher or lower concentrations will be interpreted as neurochemical modulation potentially associated with the exercise intervention and antipsychotic treatment.
  Unit: ng/mL
Serum Dopamine levels | Baseline, 12 weeks, 24 weeks, and 8-week post-intervention follow-up
  Quantification of dopamine concentration in serum using standardized laboratory procedures. Changes in dopamine concentration across timepoints will be analyzed as a marker of neurochemical modulation potentially associated with the exercise intervention and antipsychotic treatment.
  Unit: ng/mL or pg/mL

SECONDARY OUTCOMES:
Height | Baseline
  Height measured in meters using stadiometer (baseline only, if applicable)

OTHER OUTCOMES:
Sociodemographic Characterization | Baseline
  The sociodemographic characterization of participants will be performed using a structured questionnaire designed to collect information on variables such as age, gender, marital status, education, employment status, and family context. This instrument provides a comprehensive description of the sample profile and enables the analysis of potential sociodemographic factors associated with the clinical and functional variables under study.

CONTACTS AND LOCATIONS:
Locations (1):
- Local Health Unit of Trás-os-Montes and Alto Douro, Vila Real, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The dataset includes sensitive clinical, functional, and health-related information collected in a hospital setting. Data will be used exclusively for the purposes defined in the approved study protocol and in accordance with institutional ethical approval and data protection regulations.